CLINICAL TRIAL: NCT04449900
Title: Quantitative Evaluation of Parafoveal Microvasculature Changes in Eyes With Exudative Circumscribed Choroidal Haemangioma: An Optical Coherence Tomography Angiography Study
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Prof., Sun Yat-sen University
Other Study IDs: 2017MEKY034
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Circumscribed Choroidal Haemangioma; Optical Coherence Tomography Angiography; Macular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The exudative CCH group: Treatment naïve patients with exudative CCH which caused subfoveal retinal detachment and/or intraretinal fluid
  Interventions: Other: This is observational study with the examination of OCTA
- The healthy eye control group: In the healthy eye control group, all eyes should have no ocular diseases and the best-corrected visual acuity (BCVA) should be 20/20 or better.
  Interventions: Other: This is observational study with the examination of OCTA

INTERVENTIONS:
Other: This is observational study with the examination of OCTA — This is observational study with the examination of OCTA

SUMMARY:
The study aims to quantitative evaluation of parafoveal microvasculature changes in eyes with exudative circumscribed choroidal haemangioma using optical coherence tomography angiography.

DETAILED DESCRIPTION:
Circumscribed choroidal haemangioma (CCH) is an uncommon, potentially congenital benign vascular hamartomas which typically manifests as an elevated mass with reddish-orange pigmentation located posteriorly to the equator, mostly in the macular and peripapillary region. Despite its benign nature, cystoid macular edema (CME) or SRF due to the exudations from the exudative CCH can cause visual impairment. Diagnosis is often suspected clinically, and multimodal imaging is useful for the differential diagnosis of CCH from other malignant tumors such as melanoma. Optical coherence tomography angiography (OCTA) is a rapid, non-invasive, new imaging technology which could provide the capillary density (CD) of superficial and deep capillary plexus as well as the CD of choriocapillaris of the superficial, the latter two of which could not be seen on conventional FA or ICGA. However, little knowledge is known about the parafoveal microvasculature changes in eyes with exudative CCH on OCTA. Therefore, it is necessary to quantitative evaluation of parafoveal microvasculature changes in eyes with exudative CCH compared with healthy eyes without any disease. To the best of our knowledge, this is the first cross-sectional, case-control study to use OCTA to quantitative evaluation of parafoveal microvasculature changes in Eyes with exudative CCH compared with age- and gender-controlled healthy eyes.

ELIGIBILITY:
Inclusion Criteria:

* For patients with exudative CCH, the inclusion criteria were treatment naïve patients with exudative CCH which caused subfoveal retinal detachment and/or intraretinal fluid. For the healthy eye control group, only one eye (randomized by computer) of a subject was included, and the included eyes should have no ocular diseases and the best-corrected visual acuity (BCVA) should be 20/20 or better.

Exclusion Criteria:

* without any other ocular diseases or any severe uncontrolled systemic diseases, including uncontrolled hypertension, coronary heart disease, liver failure, and kidney failure. all the subjects with high diopter > -6D, long eye axis > 26.0 mm, or the quality of the acquired OCTA images below 7/10 should be excluded from this study.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: There are two groups in this study: one is the exudative CCH group,and the other is the healthy eye control group. They performed OCTA at baseline.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Quantitative changes of parafoveal microvasculature in eyes with exudative circumscribed choroidal haemangioma | 3 years
  Quantitative changes of parafoveal microvasculature in eyes with exudative circumscribed choroidal haemangioma compared wiyh healthy eyes.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No